CLINICAL TRIAL: NCT00977509
Title: Detection of Gene Mutations in Non-small Cell Lung Cancer Cells in Blood Samples or Fine-needle Aspiration
Brief Title: Gene Mutations in Non-Small Cell Lung Cancer Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812092R
Record Dates: First submitted 2009-09-10; First posted 2009-09-15 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: genes; mutation; non-small cell lung cancer; cancer cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, pleural fluid, and biopsy.
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare the frequency of individual genetic abnormality between tumor cells and blood specimens.

DETAILED DESCRIPTION:
Samples will be collected before the systemic therapy. After initiation of therapy, samples will be collected at end of the 1st month, at the end of the 2nd month at the end of 3rd months and once every three months thereafter concurrently with the tumor assessment such as time of performing CT scans. In selected consented patients, peripheral blood samples will be collected every week for the first month.

Disease status will be assessed every 2~3 months and at the end of treatment according to RECIST criteria. If progression is not observed at the end of therapy, patients will be assessed every 3 months until progression or further anti-cancer therapy. Progression-free survival, overall survival and response rate will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic or cytological confirmation of NSCLC.
* Patients must understand and provide written informed consent prior to initiation of any study-specific procedures.
* Have a life expectancy 3 months.
* Have malignant pleural/pericardial effusion or metastatic non-small cell lung cancer.
* Have measurable or evaluable disease.
* ≥20 years.
* Candidate for systemic treatment such as EGFR-TKI or chemotherapy.

Exclusion Criteria:

* Prior history of another malignancy (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study entry.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of individual genetic abnormality in advanced non-small cell lung cancer (NSCLC) patients who will commence systemic therapy. | Samples will be collected before the systemic therapy, at the end of the first three months and once every 3 months. In selected consented patients, peripheral blood samples will be collected every week for the first month.

SECONDARY OUTCOMES:
To determine the frequency with which molecular profiling of a NSCLC patient's tumor by DNA sequencing and/or FISH yields a target against which there is approved or investigational therapeutic regimen. | Samples will be collected before the systemic therapy, at the end of the first three months and once every 3 months. In selected consented patients, peripheral blood samples will be collected every week for the first month.
To determine the response rate according to RECIST, progression-free, and overall survival in patients with advanced NSCLC whose therapy is selected by molecular profile. | Disease status will be assessed every 2~3 months and at the end of treatment according to RECIST criteria. If progression is not observed at the end of therapy, patients will be assessed every 3 months until progression or further anti-cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, M.D., ph.D., Principal Investigator — National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan